CLINICAL TRIAL: NCT01102413
Title: A Phase III, Randomized, Comparative, Open-label Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by Infusions or Repeated Bolus Injections in Comparison With Oral Iron Sulphate in Subjects With Non-Dialysis Dependent Chronic Kidney Disease and With Renal-Related Anaemia
Brief Title: Iron Isomaltoside 1000 (Monofer®) in Non-Dialysis Dependent Chronic Kidney Disease and With Renal-Related Anaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-CKD-02
Record Dates: First submitted 2010-03-26; First posted 2010-04-13 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Iron Deficiency Anemia; Chronic Kidney Disease
MeSH Terms: conditions — Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monofer (Experimental): Injections or infusions
  Interventions: Drug: Monofer
- Iron Sulphate (Active Comparator): Oral intake
  Interventions: Drug: Iron Sulphate

INTERVENTIONS:
Drug: Monofer — Infusion or injections
  Arms: Monofer
Drug: Iron Sulphate — Oral intake
  Arms: Iron Sulphate

SUMMARY:
The study is designed to determine the effects of an investigational drug Monofer in subjects with non-dialysis dependent chronic kidney disease (NDD-CKD) subjects and with iron deficiency anaemia (IDA).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years.
2. Subjects diagnosed with NDD-CKD with MDRD calculated eGFR between 15-59 mL/min.
3. Hb < 11.0 g/dL (6.80 mmol/L)
4. Either or both of the following iron stores indicators below target {Serum ferritin < 100 ug/l and Transferrin saturation (TfS)<20%}.
5. Life expectancy beyond 12 months by Principal Investigator's judgement.
6. Willingness to participate after informed consent and any authorization as required by local law ( e.g. Protected Health Information [PHI] for North America).

Exclusion Criteria:

1. Anaemia predominantly caused by factors other than renal impairment or iron deficiency (according to Principal Investigator's judgment).
2. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis).
3. Drug hypersensitivity (i.e. previous hypersensitivity to Iron Dextran or iron mono- or disaccharide complexes or to iron sulphate or any excipients of the study drug.
4. Subjects with history of multiple allergies.
5. Decompensated liver cirrhosis or active hepatitis (Alanine Aminotransferase (ALT) > 3 times upper normal limit).
6. Active acute or chronic infections ((assessed by clinical judgment), supplied with White Blood Cells (WBC) and C-Reactive Protein (CRP)).
7. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
8. Pregnancy and nursing (To avoid pregnancy, women have to be postmenopausal (at least 12 months must have elapsed since last menstruation), surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product (5 days): Contraceptive pills, intrauterine devices (IUD), contraceptive depot injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches).
9. Extensive active bleeding necessitating blood transfusion.
10. Planned elective surgery during the study.
11. Participation in any other clinical study within 3 months prior to screening.
12. Known intolerance to oral iron treatment.
13. Untreated B12 or folate deficiency.
14. I.V. or oral iron treatment or blood transfusion within 4 weeks prior to screening visit.
15. ESA treatment within 8 weeks prior to screening visit.
16. Serum ferritin > 500 µg/L.
17. Any other medical condition that, in the opinion of Principal Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study or interfere with study drug evaluation. Example, Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.
18. Body weight < 30 kilograms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacosmos, Holbæk, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Monofer | Iron Sulphate
Started | 233 | 118
Completed | 208 | 106
Not Completed | 25 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monofer | Iron Sulphate | Total
Number analyzed (Participants) | 233 | 118 | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 164 | 80 | 244
  >=65 years | 69 | 38 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 54 | 195
  Male | 92 | 64 | 156
Region of Enrollment [Number; unit: participants]
  Denmark | 13 | 6 | 19
  Austria | 16 | 5 | 21
  Germany | 20 | 11 | 31
  United Kingdom | 19 | 12 | 31
  India | 138 | 64 | 202
  Poland | 4 | 4 | 8
  Russian Federation | 9 | 8 | 17
  Sweden | 1 | 0 | 1
  United States | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) Concentration From Baseline to Week 4.
Time Frame: Baseline, 4 weeks
Population: The FAS population included all the subjects who were randomised into the study, received at least one dose of the study drug, and had at least one post-baseline Hb assessment. The subjects were considered as randomised, regardless of which treatment they actually received.
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Monofer | Iron Sulphate
Number analyzed (Participants) | 209 | 108
g/dL | 0.57 [-3.1 to 4.0] | 0.35 [-3.7 to 3.9]

2. Secondary Outcome: Change in Hemoglobin Concentration From Baseline to Week 8
Time Frame: Baseline to week 8
Population: as for outcome 1
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Monofer | Iron Sulphate
Number analyzed (Participants) | 210 | 112
g/dL | 0.92 [-1.6 to 5.1] | 0.45 [-2.9 to 4.0]

ADVERSE EVENTS:
Description: The safety population included all subjects who were randomised and received at least one dose of iron isomaltoside 1000 or iron sulphate. The safety analyses was performed on the safety population.
Arm/Group | Monofer | Iron Sulphate
Serious Adverse Events (participants affected / at risk) | 12/228 | 10/117
Other Adverse Events (participants affected / at risk) | 48/228 | 22/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monofer (N=228) | Iron Sulphate (N=117)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Urinary track infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monofer (N=228) | Iron Sulphate (N=117)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 6 (7) | 1 (1)
Odema peripheral (General disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 7 (7) | 4 (4)
Nasopharyngitis (Infections and infestations) | 7 (9) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Pharmacosmos or its agents has not prepared a draft for submission to a peer reviewed journal prior to 1 year following completion of the study report, the investigators have the right to publish the results. Such publications are to be submitted to Pharmacosmos for comment 30 days prior to submision for publication.